CLINICAL TRIAL: NCT02852941
Title: Assessment of Volumetric Hemodynamic Parameters and Nutritional Status in Stable Renal Transplant Recipients
Status: Completed | Type: Observational
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Łukasz Czyżewski, PhD, Medical University of Warsaw
Other Study IDs: C.I/KTx/2016/07
Record Dates: First submitted 2016-07-27; First posted 2016-08-02 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Cardiac Output, Low; High Blood Pressure
Keywords: Impedance; Kidney Transplantation
MeSH Terms: conditions — Cardiac Output, Low; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Patients after kidney transplantation: The study included who had been admitted to a nephrology-transplantation outpatient clinic 0.5 to 30 years after kidney transplantation.
  Interventions: Device: CardioScreen 1000; Device: Tanita 418- Bioelectrical impedance analysis
- Healthy subjects: Medical staff: medical doctors, nurses
  Interventions: Device: CardioScreen 1000; Device: Tanita 418- Bioelectrical impedance analysis

INTERVENTIONS:
Device: CardioScreen 1000 — Haemodynamic Measurement System, Medis Impedance cardiography (ICG)
Device: Tanita 418- Bioelectrical impedance analysis — The device measured the size of total body water (TBW), fat mass (FM%), visceral fat%, fat free mass (FFM), and basal metabolic rate (BMR) (kcal).

SUMMARY:
Changes in volumetric hemodynamic parameters and fluid overload (Cardiac Index,Stroke Volume, Thoracic Fluid Content, Systemic Vascular Resistance) were measured using a impedance cardiography (ICG) (CardioScreen 1000 - Haemodynamic Measurement System, Medis. Ilmenau) in stable renal transplant recipients Nutritional status was measured by Tanita 418 Monitor.

ELIGIBILITY:
Inclusion Criteria:

* give voluntary consent to participate in the study
* functioning graft longer than 3 months to 10 years
* no clinical cardiovascular disease during the 6 months preceding entry
* stable graft function- glomerular filtration rate > 30 ml/min/1.73 m2, creatinine concentration <2.5 mg/dl
* medical staff (medical doctors, nurses)

Exclusion Criteria:

* not meet the above criteria
* episode of illness (for example: infection)
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 100 consecutive patients admitted to routine visin in Transplant Centre and 30 healthy subjects were included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2016-07; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Assessment of cardiac index in Stable Renal Transplant Recipients | 1 day
  Measurement of cardiac index (l/min/m2)

SECONDARY OUTCOMES:
Assessment of Nutritional Status in Stable Renal Transplant Recipients | 1 day
  Measurement of amount of fat tissue (%)
Assessment of Systemic Vascular Resistance Index in Stable Renal Transplant Recipients | 1 day
  Measurement of Systemic Vascular Resistance Index (dynes-sec/cm-5/m2)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Warsaw, Warsaw, Mazovian, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Czyzewski L, Wyzgal J, Czyzewska E, Kurowski A, Sierdzinski J, Truszewski Z, Szarpak L. Assessment of Arterial Stiffness, Volume, and Nutritional Status in Stable Renal Transplant Recipients. Medicine (Baltimore). 2016 Feb;95(6):e2819. doi: 10.1097/MD.0000000000002819. PMID 26871855
- [Background] Czyzewski L, Sanko-Resmer J, Wyzgal J, Kurowski A. Comparative analysis of hypertension and its causes among renal replacement therapy patients. Ann Transplant. 2014 Nov 3;19:556-68. doi: 10.12659/AOT.891248. PMID 25365639
- [Background] Czyzewski L, Wyzgal J, Kolek A. Evaluation of selected risk factors of cardiovascular diseases among patients after kidney transplantation, with particular focus on the role of 24-hour automatic blood pressure measurement in the diagnosis of hypertension: an introductory report. Ann Transplant. 2014 Apr 28;19:188-98. doi: 10.12659/AOT.890189. PMID 24770703
- [Background] Czyzewski L, Sanko-Resmer J, Wyzgal J, Kurowski A. Assessment of health-related quality of life of patients after kidney transplantation in comparison with hemodialysis and peritoneal dialysis. Ann Transplant. 2014 Nov 9;19:576-85. doi: 10.12659/AOT.891265. PMID 25382249